CLINICAL TRIAL: NCT00945971
Title: Catecholamine and Cognitive Response to Exercise in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Exercise Effects in Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MeirMc010-09CTIL
Record Dates: First submitted 2009-07-14; First posted 2009-07-24 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Catecholamine; Children; Physical Activity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): The intervention group will participate in an exercise program, including aerobic and anaerobic components,twice a week, for 3 months. Exercise testing, blood sampling and cognitive assessment will be performed at the start and in the end of this study.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — The intervention group will engage in exercise program, including aerobic and anaerobic components,twice a week, for 3 months. Exercise testing, blood sampling and cognitive assessment will be used at the start and in the end of this study.

SUMMARY:
The study will investigate catecholamines responses, and cognitive effects of exercise in children with attention deficit hyperactivity disorder, and the effect of exercise training on these measures.

DETAILED DESCRIPTION:
A leading pathophysiologic hypothesis of attention-deficit/hyperactivity disorder (ADHD) is based on the notion of a catecholamine [CA; norepinephrine (NE), epinephrine (EPI), and dopamine (DA)] dysfunction. This hypothesis suggests that the CA response to environmental stimuli is attenuated in ADHD and is derived primarily from observations that drugs such as methylphenidate and amphetamine - considered to be CA agonists - are effective in treating the symptoms of ADHD. Despite this compelling evidence, a definitive role of CA responsiveness in ADHD remains controversial. Physical activity is widely known to be a powerful stimulus of the hypothalamic-pituitary-adrenal (HPA) and noradrenergic systems. On the basis of the nation of a CA dysfunction in ADHD, we reasoned that the normal robust increase in circulating CA seen in response to exercise would be blunted in children with ADHD.

The objective of this study is to examine the possibility that exercise program and testing might be useful in differentiating CA responses to stress between children who had received a diagnosis of attention-deficit/hyperactivity disorder (ADHD) and age- and gender-matched controls.

This study will take place in 'Children and adolescence health and sports center' in Meir Medical Center, Kfar-Saba, Israel. Forty-five children, boys and girls between the ages 6 and 18, with newly diagnosed ADHD that not receiving any drugs will be assigned to the intervention group. Age and gender matched children with ADHD, receiving Ritalin and not engaged in regular exercise, or healthy children's without ADHD will serve as controls. The intervention group will participate in an exercise program, including aerobic and anaerobic components, twice a week, for 3 months. Exercise testing, blood sampling and cognitive assessment will be performed at the start and in the end of this study.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls between the ages 6 and 18, with newly diagnosed ADHD.

Exclusion Criteria:

* children with ADHD on medications

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Catecholamine (Epinephrine, NorEpinephrine, Dopamine) blood levels | baseline and after 3 months intervention
Exercise testing | baseline and after 3 months intervention
cognitive assessment | baseline and after 3 months intervention
  will be performed at the start and in the end of the intervention (time 0 and 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Pediatrics, Meir Medical Center, Sackler School of Medicine, Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Nemet D, Ben-Zaken S, Eliakim A. The effect of methylphenidate on the dopamine and growth hormone response to exercise in children with attention-deficit hyperactivity disorder. Growth Horm IGF Res. 2024 Jun;76:101596. doi: 10.1016/j.ghir.2024.101596. Epub 2024 May 27. PMID 38820857
- [Derived] Nemet D, Ben-Zaken S, Eliakim RA, Eliakim A. Reduced exercise-induced growth hormone secretion among children with attention-deficit hyperactivity disorder. Growth Horm IGF Res. 2022 Aug;65:101485. doi: 10.1016/j.ghir.2022.101485. Epub 2022 Jun 30. PMID 35816941